CLINICAL TRIAL: NCT06357663
Title: Effect of Subtle Energy Transmission and Tao Calligraphy Mindfulness Practice on Telomere Length in Peripheral Blood Leukocytes A Follow-up Pilot Study
Brief Title: Subtle Energy Transmission and Tao Calligraphy Mindfulness in Telomere Length in Peripheral Blood Leukocytes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This was a pilot and we achieved the goal with 12 subjects already.
Sponsor: Sha Research Foundation (Other)
Responsible Party: Principal Investigator, Peter Hudoba De Badyn MD, FRCS, Director of the Research at Sha Research Foundation, Sha Research Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00071128
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Telomere Length; Quality of Life
Keywords: Telomere Length; Leukocytes; Mindfulness; Calligraphy; Quality of Life; Tao
MeSH Terms: conditions — Thromboangiitis Obliterans

STUDY DESIGN:
Intervention Model Description: The study will be performed as a Pilot follow-up study, should the 0 Hypothesis be successfully rejected, this study will be followed by a formal Double Blind Randomized Crossover Study.
  We plan subjects may enter the study as a group and will have measurements done within short time frame from each other at beginning and at the end of 3 and 9 months.
  As this is a pilot study, there will be no randomization into treatment and control group, as a control we will use the "Normal" values of telomere from general population. All subjects will receive a transmission and then will be practicing Tao Calligraphy mindfulness daily during the 9 months.
  Every subject who is accepted into the study, will have blood sample taken for analysis and will fill Rand SF 36 Questionnaire. Afterwards, will receive transmission of subtle energy by Zhi Gang Sha (or his designee) and will be instructed on how to practice mindfulness with Tao Calligraphy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SIMPLE FOLLOW UP GROUP (Other): Every subject who is accepted into the study, will receive prior to the inception of practice transmission of pure energy (blessing) and will be instructed on how to practice meditations with Tao Calligraphy.
  Blood samples will be drawn at DAP accredited institution in British Columbia (Life Labs or Vancouver Coastal Health) and will be promptly sent by currier to Repeat Diagnostics, All participants will have blood samples drawn and Questionnaire filled at the entry time point (Time 0), at the end of 3 months (Time 1), and at the end of 9 months (Time 2).
  Interventions: Other: Mindfulness practice with Calligraphy

INTERVENTIONS:
Other: Mindfulness practice with Calligraphy — The unique style of Art Meditation where mindfulness (heightened awareness) is achieved by combination of movement and focus on Chinese Tao Calligraphy while chanting a mantra. The practitioners repeatedly trace the lines of Tao calligraphy with fingers and chant the mantra. This enables them to achieve deep concentration, while maintaining fully alert state. The practice can be done in sitting or standing, depending on the health status and age.

SUMMARY:
Effect of Subtle Energy Transmission and Tao Calligraphy Mindfulness Practice on Telomere Length in Peripheral Blood Leukocytes A Follow-up Pilot Study

The goal of this Pilot clinical trial is to learn if a Subtle Energy Transmission and Tao Calligraphy Mindfulness Practice works to increase Telomere Length in Peripheral Blood Leukocytes in adults. The main questions it aims to answer are:

* Does A Subtle energy transmission and Tao Calligraphy Mindfulness increase Telomere Length in Peripheral Blood Leukocytes in adults?
* Will this increase of Telomere Length in Peripheral Blood Leukocytes in adults be statistically significant? Researchers will compare the length of Telomere in peripheral blood Leukocytes at beginning of the mindfulness practices to the length of Telomere in peripheral blood Leukocytes at 3 months and at 9 months of regular daily practices.

Participants will:

* Receive a transmission of Subtle energy at beginning of practices
* Visit the Laboratory for a blood sample taken at beginning, at 3 months and at 9 months of practices.
* Fill the Study Questionnaires at beginning, at 3 months and at 9 months of practices.
* Practice the Mindfulness with Tao Calligraphy daily 1 hour in the morning and 1 hour in the evening.

DETAILED DESCRIPTION:
OBJECTIVES The proposed research is a pilot project based on experiential data obtained from several previous pilot and formal studies by the investigators' research teams and by researchers from other institutions. It is intended to measure the effects of the transmission of subtle energy (blessing), combined with a specific form of meditation, on the length of human telomeres in peripheral blood leucocytes and on overall well-being. The investigators hope that the study will provide further data for individuals seeking an additional modality to prolong life expectancy that could be integrated into conventional medical protocols.

HYPOTHESIS The research null hypothesis is that individuals who receive a subtle energy transmission for improving telomere length in peripheral blood leucocytes and who will also then regularly practice mindfulness with Tao Calligraphy for nine months will (a) have no significant change in telomere length in follow-up analyses as measured by telomere length in peripheral blood leukocytes and will (b) show no improvement of well-being as assessed via the standardized scientific questionnaire Rand SF 36(s) at three and nine months.

Statistical test Anova (using Minitab version 14 and PSPP/SPSS) will be used to evaluate the null hypothesis. The p-value will represent how unlikely the observed data would be if the null hypothesis were actually true and the investigators will use them to reach conclusions. The investigators set the confidence level at 95% and if p <= 0.05, then H0 is rejected.

BACKGROUND Telomeres as Markers of Longevity Background: Telomeres are distinctive protein-DNA structures (repetitive (TTAGGG) sequences) at the end of the chromosomes that are essential for maintaining the integrity and stability of the genome. Telomere length shortens with age (due to multiple cell divisions). The rate of telomere shortening has been found to increase or decrease in association with specific lifestyle factors.

To counteract the loss of telomere repeats with each cell division, germline cells, highly proliferating cells from the skin, the gut, and hematopoietic tissues, as well as tumor cells, express DNAmAge telomerase, an enzyme complex with reverse transcriptase activity, which adds the necessary telomeric DNA (T2AG3 repeats) to the 3-end of the telomeres, protecting their degeneration. Despite expression of telomerase, the telomere length in highly proliferating cells from long-lived species decreases during development and with replication in vitro and with age in vivo. Most likely, telomerase levels in such cells are tightly regulated and are insufficient to make up for the net loss of telomere repeats with cell division.

The telomere length values reflect telomere shortening (resulting from cell divisions, oxidative damage, and other causes) and telomere elongation (mainly resulting from telomerase activity) of the chromosome-specific telomere length inherited in the gametes. Consequently, researchers have two main tools to analyze telomeres, the telomere length and the telomerase.

Although the ability of telomere length measured in peripheral blood to predict life expectancy or monitor mechanisms underlying the aging process is not entirely consistent across studies, telomere length currently remains one of the most widely used biomarkers in epidemiological and clinical studies of aging.

In the protocol of the study, the investigators have discussed several studies using either of these two markers.

The laboratory test used in this study to measure telomere length The average length of telomere repeats can be measured by in situ hybridization and flow cytometry [flow-FISH]. In order to measure the telomere length in granulocytes, naive T cells, memory T cells, B cells, and natural killer (NK)/NKT cells within a blood sample, flow-FISH can be combined with antibody-staining (Multicolor flow-FISH). Most steps in the staining protocol are automated using a 96-well micro-dispenser device. The minimum detectable difference in telomere length and the reproducibility of the method are in the range of 0.2-0.5 kb and measurements can be made with as few as a thousand cells. Automated multicolor flow-FISH greatly facilitates studies of telomere length regulation in subsets of nucleated blood cells, especially when only few cells are available and when differences in telomere length are small.

In Repeat Diagnostics, the laboratory being used for this study, the fluorescent signals from telomeres are assessed on a single cell basis by flow cytometry, with patient results reported for lymphocytes, granulocytes, B-cells, naïve and memory T-cells, and NK cells. All patient telomere length profiles are reported in relationship to age-matched controls and are available for all age ranges from pediatric to geriatric. This telomere reference curve was established by the study of over 800 healthy individuals between birth and 100 years of age. This informative technique allows analysis and comparisons of the telomere length between different cell types and within one cell type, e.g., in differentiating between constitutional deficiencies and specific cell type deficiencies.

The test used in this study to measure overall effect of mindfulness practice A 36-item short-form Quality of Life Questionnaire (SF-36) was constructed to survey health status in the Medical Outcomes Study. The SF-36 was designed for use in clinical practice and research, health policy evaluations, and general population surveys. Although the 12-item short-form of SF-36 would be easier to use, the investigators chose the longer 36-item version, as standard errors were described nearly always to be larger for the 12-item short-form.

The SF-36 includes one multi-item scale that assesses eight health concepts:

1. limitations in physical activities because of health problems;
2. limitations in social activities because of physical or emotional problems;
3. limitations in usual role activities because of physical health problems;
4. bodily pain;
5. general mental health (psychological distress and well-being);
6. limitations in usual role activities because of emotional problems;
7. vitality (energy and fatigue); and
8. general health perceptions.

Through a complex calculation, eight scores are derived from answers to 36 questions of SF-36. Finally, these eight scores are linearly transformed to a 0-to-100 scale, with 100 being the best possible outcome.

Chinese calligraphy Chinese calligraphic writing uses an ink-laden brush to create defined configurations of characters. Studies of Chinese calligraphic writing have confirmed its significant effects on psychosomatic conditions, post-traumatic hyper-arousal symptoms, hypertension, and type 2 diabetes.

The investigators chose a Tao Calligraphy practice, which is unique style of moving meditation, wherein mindfulness (heightened awareness) is achieved by the combination of movement and focus on a work of Tao Calligraphy art. In this practice, the subjects do not use an ink-laden brush to write on the paper, but trace the strokes of premade calligraphy with fingers and simultaneously repeat an affirmation (mantra) aloud or silently, which enables them to achieve deep concentration during wakefulness.

Results from the investigators of previous studies confirmed the efficacy of this practice, with significant results in improving overall well-being and chronic conditions as documented by SF MPQ (McGill Pain Questionnaire), by EORTC QLQ-30 (Cancer Quality of Life Questionnaire), and by SF-36 (Quality of Life Questionnaire).

METHOD The study will be performed as a pilot follow-up study. Should the null hypothesis be successfully rejected, this study will be followed by a formal Double Blind Randomized Crossover Study.

As this is a pilot study, there will be no randomization into intervention and control groups. As a control, the investigators will use the "normal" values from the general population. All subjects will receive a transmission and then will be practicing Tao Calligraphy mindfulness daily during the nine-month duration of the study.

The study is conducted on an outpatient basis and includes:

* Informational telephone or Zoom meeting to clarify inclusion/exclusion criteria, the study design, and the consent/information forms, with signing thereof
* Initial instructional Zoom meeting to teach the practice of Tao Calligraphy tracing meditation and to deliver the subtle energy transmission (blessing)
* Laboratory assessment of telomere length in peripheral blood leucocytes of participants
* Completion of the questionnaires by participants
* Completion of assessments by a study principal and co-investigators

Laboratory assessment of telomere length in peripheral blood leucocytes:

Laboratory assessment of telomere length in peripheral blood leucocytes will be performed at the entry time point (Time 0), at the end of three months (Time 1), and at the end of nine months (Time 2) for every participant.

Blood samples will be drawn at "Life Labs," a DAP-accredited institution in British Columbia and an accredited institution in the United States, and will be promptly sent by courier to Repeat Diagnostics, Suite 309 - 267 West Esplanade, North Vancouver, BC V7M 1A5 Canada for telomere assessment by Flow FISH.

Reports will be issued to clinical Principal Investigator, Dr. Peter Hudoba.

Improvement of general well-being or clinical well-being as measured by standardized questionnaires:

1. John Ware's SF-36 Quality of Life questionnaire
2. Simple follow-up questionnaire of the investigators' own design (to address any additional information participants may have).

Participants will complete both questionnaires online on the Sha Research Foundation website using unique IDs to secure confidentiality.

Each subject of the study will answer all 36 questions at the entry time point (Time 0), at the end of three months (Time 1), and at the end of nine months (Time 2).

From the SF-36 answers, the study statistician will derive 8 scores in a blind fashion. Then, the 8 scores from beginning and end data will be compared to each other and to "normal" values using Anova test. As a control, the investigators will use "normal" values corresponding to the age of each participant at the beginning and at the end of their participation.

The correlation coefficient will be used to determine any correlations between various factors (e.g., effects of age, sex, length, frequency of mindfulness practices, and others) on outcomes and regression analysis to determine the relationship between independent and dependent variables.

Data will be stored on an external hard drive to prevent unauthorized access through the internet.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects / patients (age 60 years and over) we expect at 60 years people have already measurable shortening of telomeres
* Healthy or Ill, with the exception of genetic illnesses and cancer (for which treatments could negatively impact telomeres)
* Willingness and ability to comply with data collection requirements.
* Complete submission of required documentation prior to enrollment into the study, including informed consent and consent to release of information.
* Willingness to allow their data to be used for research purposes and published as deemed fit (while conforming to all applicable privacy laws) by Sha Research Foundation.
* Willingness to practice the daily calligraphy meditations and follow the protocol.

Exclusion Criteria:

* Not meeting any of the inclusion criteria
* Bipolar disorders, other serious mental disorders (e.g. schizophrenia, psychosis), genetic illnesses (primarily affected chromosomes), and cancer (treatment could negatively impact telomere during research period)
* inability to sign consent and follow instructions
* Unwillingness to participate in data gathering
* Unable to follow the practice regimen, including the daily calligraphy meditations
* Pregnant or nursing. Participants who become pregnant during the study will be required to end their participation. (to avoid any, at current time unknown, potential negative effect of the study on the fetus).
* There are no exclusion criteria placed upon potential subjects related to national origin, culture, ethnicity, race, sex, physical disability, sexual orientation, religion, or spiritual practices.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Telomere Length in Peripheral blood leukocytes | 9 months
  The Change of Telomere Length in Peripheral blood leukocytes after 9 months of Mindfulness Practice with Tao Calligraphy

SECONDARY OUTCOMES:
Quality of Life by John Ware's SF-36 Quality of Life questionnaire (that produces eight scores with 0-to-100 scale, 100 being the best possible outcome). | 9 months
  The Change of Quality of Life by John Ware's SF-36 Quality of Life questionnaire after 9 months of Mindfulness Practice with Tao Calligraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hudoba De Badyn, MD, FRCS, Principal Investigator — Sha Research Foundation
Locations (1):
- Sha Research Foundation (Branch), North Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Will need to contact IRB if permitted, as this is not in approved protocol
Supporting Information: Study Protocol, SAP
Time Frame: September 2024 to March 2025
Access Criteria: Anyone on Clinical Trials Gov

REFERENCES:
- [Background] Jacobs TL, Epel ES, Lin J, Blackburn EH, Wolkowitz OM, Bridwell DA, Zanesco AP, Aichele SR, Sahdra BK, MacLean KA, King BG, Shaver PR, Rosenberg EL, Ferrer E, Wallace BA, Saron CD. Intensive meditation training, immune cell telomerase activity, and psychological mediators. Psychoneuroendocrinology. 2011 Jun;36(5):664-81. doi: 10.1016/j.psyneuen.2010.09.010. Epub 2010 Oct 29. PMID 21035949
- [Background] Dal Lin C, Marinova M, Brugnolo L, Rubino G, Plebani M, Iliceto S, Tona F. Rapid changes of miRNAs-20, -30, -410, -515, -134, and -183 and telomerase with psychological activity: A one year study on the relaxation response and epistemological considerations. J Tradit Complement Med. 2021 Feb 15;11(5):409-418. doi: 10.1016/j.jtcme.2021.02.005. eCollection 2021 Sep. PMID 34522635
- [Background] Pavanello S, Campisi M, Tona F, Lin CD, Iliceto S. Exploring Epigenetic Age in Response to Intensive Relaxing Training: A Pilot Study to Slow Down Biological Age. Int J Environ Res Public Health. 2019 Aug 23;16(17):3074. doi: 10.3390/ijerph16173074. PMID 31450859
- [Background] Thimmapuram J, Pargament R, Sibliss K, Grim R, Risques R, Toorens E. Effect of heartfulness meditation on burnout, emotional wellness, and telomere length in health care professionals. J Community Hosp Intern Med Perspect. 2017 Mar 31;7(1):21-27. doi: 10.1080/20009666.2016.1270806. eCollection 2017 Jan. PMID 28634520
- [Background] Liu Z, Kuo PL, Horvath S, Crimmins E, Ferrucci L, Levine M. Correction: A new aging measure captures morbidity and mortality risk across diverse subpopulations from NHANES IV: A cohort study. PLoS Med. 2019 Feb 25;16(2):e1002760. doi: 10.1371/journal.pmed.1002760. eCollection 2019 Feb. PMID 30802240
- [Background] Liu Z, Kuo PL, Horvath S, Crimmins E, Ferrucci L, Levine M. A new aging measure captures morbidity and mortality risk across diverse subpopulations from NHANES IV: A cohort study. PLoS Med. 2018 Dec 31;15(12):e1002718. doi: 10.1371/journal.pmed.1002718. eCollection 2018 Dec. PMID 30596641
- [Background] Lu AT, Quach A, Wilson JG, Reiner AP, Aviv A, Raj K, Hou L, Baccarelli AA, Li Y, Stewart JD, Whitsel EA, Assimes TL, Ferrucci L, Horvath S. DNA methylation GrimAge strongly predicts lifespan and healthspan. Aging (Albany NY). 2019 Jan 21;11(2):303-327. doi: 10.18632/aging.101684. PMID 30669119
- [Background] Field AE, Robertson NA, Wang T, Havas A, Ideker T, Adams PD. DNA Methylation Clocks in Aging: Categories, Causes, and Consequences. Mol Cell. 2018 Sep 20;71(6):882-895. doi: 10.1016/j.molcel.2018.08.008. PMID 30241605
- [Background] Goldman EA, Eick GN, Compton D, Kowal P, Snodgrass JJ, Eisenberg DTA, Sterner KN. Evaluating minimally invasive sample collection methods for telomere length measurement. Am J Hum Biol. 2018 Jan;30(1):10.1002/ajhb.23062. doi: 10.1002/ajhb.23062. Epub 2017 Sep 26. PMID 28949426
- [Background] Ahadi S, Zhou W, Schussler-Fiorenza Rose SM, Sailani MR, Contrepois K, Avina M, Ashland M, Brunet A, Snyder M. Personal aging markers and ageotypes revealed by deep longitudinal profiling. Nat Med. 2020 Jan;26(1):83-90. doi: 10.1038/s41591-019-0719-5. Epub 2020 Jan 13. PMID 31932806
- [Background] Gorenjak V, Akbar S, Stathopoulou MG, Visvikis-Siest S. The future of telomere length in personalized medicine. Front Biosci (Landmark Ed). 2018 Mar 1;23(9):1628-1654. doi: 10.2741/4664. PMID 29293454
- [Background] Notterman DA, Schneper L. Telomere Time-Why We Should Treat Biological Age Cautiously. JAMA Netw Open. 2020 May 1;3(5):e204352. doi: 10.1001/jamanetworkopen.2020.4352. No abstract available. PMID 32364591
- [Background] Koliada AK, Krasnenkov DS, Vaiserman AM. Telomeric aging: mitotic clock or stress indicator? Front Genet. 2015 Mar 16;6:82. doi: 10.3389/fgene.2015.00082. eCollection 2015. No abstract available. PMID 25852738
- [Background] Sanders JL, Newman AB. Telomere length in epidemiology: a biomarker of aging, age-related disease, both, or neither? Epidemiol Rev. 2013;35(1):112-31. doi: 10.1093/epirev/mxs008. Epub 2013 Jan 9. PMID 23302541
- [Background] Vaiserman A, Krasnienkov D. Telomere Length as a Marker of Biological Age: State-of-the-Art, Open Issues, and Future Perspectives. Front Genet. 2021 Jan 21;11:630186. doi: 10.3389/fgene.2020.630186. eCollection 2020. PMID 33552142
- [Background] Skytthe A, Pedersen NL, Kaprio J, Stazi MA, Hjelmborg JV, Iachine I, Vaupel JW, Christensen K. Longevity studies in GenomEUtwin. Twin Res. 2003 Oct;6(5):448-54. doi: 10.1375/136905203770326457. PMID 14624729
- [Background] Herskind AM, McGue M, Holm NV, Sorensen TI, Harvald B, Vaupel JW. The heritability of human longevity: a population-based study of 2872 Danish twin pairs born 1870-1900. Hum Genet. 1996 Mar;97(3):319-23. doi: 10.1007/BF02185763. PMID 8786073
- [Background] vB Hjelmborg J, Iachine I, Skytthe A, Vaupel JW, McGue M, Koskenvuo M, Kaprio J, Pedersen NL, Christensen K. Genetic influence on human lifespan and longevity. Hum Genet. 2006 Apr;119(3):312-21. doi: 10.1007/s00439-006-0144-y. Epub 2006 Feb 4. PMID 16463022
- [Background] Boyce WT, Sokolowski MB, Robinson GE. Genes and environments, development and time. Proc Natl Acad Sci U S A. 2020 Sep 22;117(38):23235-23241. doi: 10.1073/pnas.2016710117. PMID 32967067
- [Background] Steenman M, Lande G. Cardiac aging and heart disease in humans. Biophys Rev. 2017 Apr;9(2):131-137. doi: 10.1007/s12551-017-0255-9. Epub 2017 Mar 20. PMID 28510085
- [Background] Kalyani RR, Egan JM. Diabetes and altered glucose metabolism with aging. Endocrinol Metab Clin North Am. 2013 Jun;42(2):333-47. doi: 10.1016/j.ecl.2013.02.010. Epub 2013 Mar 22. PMID 23702405
- [Background] Aunan JR, Cho WC, Soreide K. The Biology of Aging and Cancer: A Brief Overview of Shared and Divergent Molecular Hallmarks. Aging Dis. 2017 Oct 1;8(5):628-642. doi: 10.14336/AD.2017.0103. eCollection 2017 Oct. PMID 28966806
- [Background] Kao H Sr, Zhu L, Chao AA, Chen HY, Liu IC, Zhang M. Calligraphy and meditation for stress reduction: an experimental comparison. Psychol Res Behav Manag. 2014 Feb 13;7:47-52. doi: 10.2147/PRBM.S55743. eCollection 2014. PMID 24611024
- [Background] Kao HS, Lam SP, Kao TT. Chinese calligraphy handwriting (CCH): a case of rehabilitative awakening of a coma patient after stroke. Neuropsychiatr Dis Treat. 2018 Jan 31;14:407-417. doi: 10.2147/NDT.S147753. eCollection 2018. PMID 29440902
- [Background] Zhu Z, Wang R, Kao HS, Zong Y, Liu Z, Tang S, Xu M, Liu IC, Lam SP. Effect of calligraphy training on hyperarousal symptoms for childhood survivors of the 2008 China earthquakes. Neuropsychiatr Dis Treat. 2014 Jun 3;10:977-85. doi: 10.2147/NDT.S55016. eCollection 2014. PMID 24940061
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ware JE Jr. SF-36 health survey update. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3130-9. doi: 10.1097/00007632-200012150-00008. No abstract available. PMID 11124729
- [Background] Baerlocher GM, Lansdorp PM. Telomere length measurements in leukocyte subsets by automated multicolor flow-FISH. Cytometry A. 2003 Sep;55(1):1-6. doi: 10.1002/cyto.a.10064. PMID 12938182
- Available data/document: Study Protocol: Pro00071128 — https://www.advarra.com/review-services/institutional-review-board/canadian-review-services/ — Upon request, ADVARRA (IRB) can provide your with Study Protocol + Statistical Plan, Informed Consent Form, and any other reviewed and approved documents of the study. Should you require any more information, please contact me on email sharesearchfoundation@yahoo.ca and I will provide you with any documents relevant to the study. Peter Hudoba De Badyn FRCS

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT06357663/Prot_SAP_000.pdf